CLINICAL TRIAL: NCT03773757
Title: Indiana Palliative Excellence in Alzheimer's Care Efforts- Randomized Control Trial
Brief Title: Indiana Palliative Excellence in Alzheimer's Care Efforts
Acronym: IN-PEACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Regenstrief Institute, Inc. (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Greg Sachs, Professor of Medicine, Division Chief General Internal Medicine and Geriatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1707549593; 1R01AG057733-01A1 (NIH)
Record Dates: First submitted 2018-11-21; First posted 2018-12-12 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IN-PEACE Dementia Care Coordination (Experimental): In-PEACE intervention arm will have monthly contact with a dementia care coordinator (DCC) to to identify symptoms the person with memory problems is having, including: pain, sadness, or other symptoms. The Dementia Care Coordinator will consult with the project clinical team to develop a plan of care utilizing standardized protocols to reduce the burdens of disease associated symptoms and behaviors.
  Interventions: Behavioral: IN-PEACE Dementia Care Coordination
- Usual Care (No Intervention): The usual care arm will have access to education and informational materials from the local chapter of the Alzheimer's Association and other community resources and will be reminded of these resources throughout the study.

INTERVENTIONS:
Behavioral: IN-PEACE Dementia Care Coordination — Patient/Caregivers assigned to the intervention arm will have monthly phone calls with a Nurse or Social Worker, in the capacity of a Dementia care coordinator (DCC) to identify symptoms and behavior problems the person with memory problems is having, including: pain, sadness, or other symptoms. The Dementia Care Coordinator will consult with the project clinical team to develop a plan of care utilizing standardized protocols to reduce the burdens of disease associated symptoms and behaviors. In addition, education and support materials will be provided to the caregiver in the role caring and management of a patient with dementia.
  Arms: IN-PEACE Dementia Care Coordination

SUMMARY:
The overarching goal of this research is to improve the care of community dwelling patients with dementia and their family caregivers through an innovative model of supportive care that combines an existing, evidence-based intervention for dementia care with an innovative intervention for palliative care in dementia. The intervention projects this care into the homes of patients and caregivers, empowering caregivers, and integrating with ongoing care. IN-PEACE will enroll 200 patient-caregiver dyads, randomizing 100 dyads each to the intervention and usual care arms and follow for 24 months with quarterly outcome assessments. The core of the multi-component intervention is regular, proactive telephone contact by a dementia care coordinator (DCC; social worker or RN) to anticipate and identify patients' symptoms and caregivers needs and address by utilizing specific, evidence-based protocols. Protocols cover basic dementia care, caregiver distress, neuropsychiatric symptoms, pain, navigating the hospital, feeding difficulties, and transition to hospice. The intervention also involves advance care planning and support with caregivers tailored to decisions faced in dementia care, highlighting where palliative care options can replace the default that often results in burdensome treatments.

The primary aim of IN-PEACE is to test the effect of the intervention on patients' neuropsychiatric symptoms. Other aims include testing the effect of IN-PEACE on patients' overall symptom outcomes, caregiver mood and distress, and the provision of burdensome treatments to patients (hospitalizations and emergency room visits).

DETAILED DESCRIPTION:
Dementia is an increasingly prevalent, costly and burdensome condition. The dramatic aging of the US population is creating a dementia "epidemic" that our health care system is poorly prepared to handle. More than 5 million people are affected by Alzheimer's disease (AD) and related dementias in 2016, with that number estimated to nearly triple to 13.8 million by 2050. The direct health care costs alone for dementia care are projected to increase from $236 billion in 2016 to more than $1 trillion in 2050. In addition to cognitive and functional deterioration, patients with dementia experience behavioral and psychological complications such as agitation and depression. Family caregivers of patients with dementia experience higher levels of anxiety, depression, chronic fatigue, and an increased mortality risk.

Dementia and palliative care are national research priorities. Both dementia and palliative care have been identified as priority conditions for research and quality improvement by numerous organizations such as the Institute of Medicine, National Quality Forum, the Centers for Medicare and Medicaid Services, and Agency for Healthcare Research and Quality and National Institute on Aging. In addition, a workgroup developing milestones for care and support under the U.S. National Alzheimer's Plan has explicitly stated that palliative care needs to be incorporated throughout the course of caring for patients and families affected by dementia.

2.0 Rationale and Specific Aims

Aim 1: To test the effect of the IN-PEACE intervention on patients' neuropsychiatric symptoms (e.g., agitation/aggression, anxiety, repetitive behaviors). Mixed effects models will be used to compare repeated Neuropsychiatric Inventory Questionnaire (NPI-Q) scores obtained at 3, 6, 9, 12, 15, 18, 21, and 24 months. Repeatedly measured NPI-Q scores will be the dependent variable in the model.

Aim 2: To test the effect of the IN-PEACE intervention on patients' overall symptom outcomes. Analyses in this aim will use repeatedly measured Symptom Measures in End-of-Life Dementia (SM-EOLD) scores over 24 months of follow-up as the dependent variable in the mixed effects model, similarly to the approach described for Aim 1.

Aim 3: To test the effect of the IN-PEACE intervention on caregivers' distress and mood. Aim 3 analyses will use repeatedly measured caregiver NPI-Q distress scores and caregiver Patient Health Questionnaire (PHQ-9) over 24 months of follow-up as the dependent variables in separate mixed effects models, similar to the approach for Aim 1.

Aim 4: Evaluate the effect of the IN-PEACE intervention on ER/hospital use. ER/hospitalization events will be obtained from accessing electronic medical records maintained by the Indiana Health Information Exchange (IHIE) and the Indiana Network for Patient Care (INPC). Poisson regression models will be used to compare rates of any ER/hospitalization event between the two groups while adjusting for dementia severity and significant baseline variables that differ between the two groups.

ELIGIBILITY:
Inclusion Criteria: Community-dwelling and living in the Indianapolis metropolitan area; Patient with an established diagnosis of dementia of any etiology; Dementia in the moderate (FAST stage 5) to severe stage (FAST 6-7); and English-speaking Primary caregiver informant enrolled in study.

Exclusion Criteria: Patient with dementia residing in a nursing facility or receiving hospice care; Patient or Caregiver with long-standing history of severe mental illness or Psychiatric disorder preexisting the dementia diagnosis. Initially, non-English speaking patients were excluded. On April 14, 2020, Institutional Review Board (IRB) Amendment eliminated this exclusion so non-English speaking patients could be enrolled as long as their Caregiver was English-speaking and able to complete assessments.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 402 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2023-01-07 (Actual); Study Completion 2023-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg A Sachs, MD, Principal Investigator — Indiana University
Locations (1):
- Sandra Eskenazi Center for Brain Care Innovation, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kaufer DI, Cummings JL, Ketchel P, Smith V, MacMillan A, Shelley T, Lopez OL, DeKosky ST. Validation of the NPI-Q, a brief clinical form of the Neuropsychiatric Inventory. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):233-9. doi: 10.1176/jnp.12.2.233. PMID 11001602
- [Result] Volicer L, Hurley AC, Blasi ZV. Scales for evaluation of End-of-Life Care in Dementia. Alzheimer Dis Assoc Disord. 2001 Oct-Dec;15(4):194-200. doi: 10.1097/00002093-200110000-00005. PMID 11723370
- [Result] Lowe B, Unutzer J, Callahan CM, Perkins AJ, Kroenke K. Monitoring depression treatment outcomes with the patient health questionnaire-9. Med Care. 2004 Dec;42(12):1194-201. doi: 10.1097/00005650-200412000-00006. PMID 15550799
- [Derived] Sachs GA, Johnson NM, Gao S, Torke AM, Hickman SE, Pemberton A, Vrobel A, Pan M, West J, Kroenke K. Palliative Care Program for Community-Dwelling Individuals With Dementia and Caregivers: The IN-PEACE Randomized Clinical Trial. JAMA. 2025 Mar 18;333(11):962-971. doi: 10.1001/jama.2024.25845. PMID 39878993
- [Derived] Holtz LR, Kroenke K, Gao S, Hickman SE, Torke AM, Johnson NM, Pemberton A, Vrobel A, Pan M, Sachs GA. Indiana Palliative Excellence in Alzheimer's Care Efforts (IN-PEACE): Protocol for a randomized controlled trial in persons with advanced dementia. Contemp Clin Trials. 2023 Jul;130:107217. doi: 10.1016/j.cct.2023.107217. Epub 2023 May 4. PMID 37149000

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on 3/14/2019 and ended on 12/21/2020. Recruitment locations included two health systems and personal referrals at a caregiver symposium within a 50-mile radius of Indianapolis. Initially, recruitment included an in-person approach in the medical clinic followed by in-person enrollment in the caregiver's home. After the Institutional Review Board (IRB) approved verbal consent 3/17/2020, all recruitment took place over the phone.
Pre-assignment Details: Data values reported in the Participant Flow represent individual participants.
Period: Overall Study
Arm/Group | IN-PEACE Dementia Care Coordination | Usual Care
Started | 198 | 204
Completed | 196 | 200
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Population: These variables were collected for all participant dyads (patient plus caregiver) randomized to either the usual care arm or dementia care coordination arm. Some variables may not total overall participants if caregiver opted not to answer that item.
Units Other Than Participants: Dyad: Patient and Caregiver
Groups:
- Total: Total of all reporting groups
Arm/Group | IN-PEACE Dementia Care Coordination | Usual Care | Total
Number analyzed (Participants) | 99 | 102 | 201
Number analyzed (Dyad: Patient and Caregiver) | 99 | 102 | 201
Age, Continuous [Mean (Standard Deviation); unit: years]
  Patient Participants | 83.7 (7.7) | 83.4 (8.1) | 83.6 (7.9)
  Caregiver Participants | 60.8 (12.3) | 60.2 (10.1) | 60.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Patient Participants: Female | 67 | 69 | 136
  Patient Participants: Male | 32 | 33 | 65
  Caregiver Participants: Female | 82 | 81 | 163
  Caregiver Participants: Male | 17 | 21 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — During baseline, the question was asked: What ethnic group would you consider yourself to be a member? Responses available were: Hispanic or Latino, Not Hispanic or Latino, or Refused to answer.
  Participants
    Patient Participants: Hispanic or Latino | 2 | 3 | 5
    Patient Participants: Not Hispanic or Latino | 94 | 95 | 189
    Patient Participants: Unknown or Not Reported | 3 | 4 | 7
    Caregiver Participants: Hispanic or Latino | 2 | 3 | 5
    Caregiver Participants: Not Hispanic or Latino | 94 | 94 | 188
    Caregiver Participants: Unknown or Not Reported | 3 | 5 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Caregivers chose 1 or more options for race for themselves and the person with dementia (PWD): American Indian or Alaskan Native, Asian, Pacific Islander, African American (not Hispanic), Filipino, White or Refused to answer. To ensure statistical power for analyses, those who chose African American as at least one race they identified with are counted as African American. Other combinations not included in African American or White are counted as Others.
  Participants
    African American: PWD | 44 | 43 | 87
    African American: Caregiver | 43 | 46 | 89
    White: PWD | 48 | 53 | 101
    White: Caregiver | 49 | 52 | 101
    Others: PWD | 3 | 4 | 7
    Others: Caregiver | 3 | 2 | 5
    Refused to Answer: PWD | 4 | 2 | 6
    Refused to Answer: Caregiver | 4 | 2 | 6
Region of Enrollment [Number; unit: Dyad: Patient and Caregiver] — All dyads (patient and caregiver) were enrolled within 50-mile radius of metropolitan Indianapolis, Indiana area.
  Dyad: Patient and Caregiver
    United States | 99 | 102 | 201
Education [Count of Participants; unit: Participants] — Caregivers were asked to identify their own education level and the education level of the person with dementia (PWD): high school or less, some college or college degree, post graduate.
  Participants
    PWD: High School or Less | 53 | 53 | 106
    PWD: Some college or college degree | 30 | 29 | 59
    PWD: Post graduate | 16 | 19 | 35
    PWD: did not answer | 0 | 1 | 1
    Caregiver: High School or Less | 13 | 18 | 31
    Caregiver: Some college or college degree | 60 | 54 | 114
    Caregiver: Post graduate | 26 | 29 | 55
    Caregiver: did not answer | 0 | 1 | 1
Marital Status [Count of Participants; unit: Participants] — Caregivers chose marital status for themselves and for person with dementia (PWD): Single never married, Married, Widowed, Divorced, Separated, or Living together.
  Participants
    PWD: Divorced/Separated | 25 | 12 | 37
    PWD: Married/Living together | 32 | 30 | 62
    PWD: Never Married | 6 | 8 | 14
    PWD: Widowed | 36 | 52 | 88
    Caregiver: Divorced/Separated | 13 | 15 | 28
    Caregiver: Married/Living together | 66 | 71 | 137
    Caregiver: Never Married | 19 | 13 | 32
    Caregiver: Widowed | 1 | 3 | 4
Income [Count of Participants; unit: Participants] — Caregivers chose income range for themselves as well as the person with dementia (PWD): under $24,999, $25,000-49,999, $50,000-99,999, $100,000 and over, do not wish to answer.
  If the caregiver relationship to the PWD was spouse, then the income range chosen for the caregiver counted as that of the PWD.
  Participants
    PWD : Under $24,999: Yes | 46 | 37 | 83
    PWD : Under $24,999: No | 53 | 65 | 118
    PWD : $25,000 - 49,999: Yes | 12 | 21 | 33
    PWD : $25,000 - 49,999: No | 87 | 81 | 168
    PWD : $50,000 - 99,999: Yes | 6 | 7 | 13
    PWD : $50,000 - 99,999: No | 93 | 95 | 188
    PWD : $100,000 and over: Yes | 3 | 5 | 8
    PWD : $100,000 and over: No | 96 | 97 | 193
    PWD : Do not wish to answer: Yes | 10 | 14 | 24
    PWD : Do not wish to answer: No | 89 | 88 | 177
    PWD : Caregiver is the spouse: Yes | 20 | 18 | 38
    PWD : Caregiver is the spouse: No | 79 | 84 | 163
    Caregiver : Under $24,999: Yes | 13 | 13 | 26
    Caregiver : Under $24,999: No | 86 | 89 | 175
    Caregiver : $25,000 - 49,999: Yes | 26 | 29 | 55
    Caregiver : $25,000 - 49,999: No | 73 | 73 | 146
    Caregiver : $50,000 - 99,999: Yes | 23 | 21 | 44
    Caregiver : $50,000 - 99,999: No | 76 | 81 | 157
    Caregiver : $100,000 and over: Yes | 24 | 29 | 53
    Caregiver : $100,000 and over: No | 75 | 73 | 148
    Caregiver : Do not wish to answer: Yes | 13 | 10 | 23
    Caregiver : Do not wish to answer: No | 86 | 92 | 178
Caregiver Relationship to Patient [Count of Participants; unit: Participants] — Caregivers identified their relationship to the person with dementia (PWD): spouse/partner, daughter/son/daughter-in-law/son-in-law, grandchild, or other relationship.
  Participants
    Spouse/Partner | 22 | 22 | 44
    Daughter/Son/Daughter-in-Law/Son-in-Law | 68 | 67 | 135
    Grandchild | 1 | 2 | 3
    Other relationship | 8 | 11 | 19
Patient Institution [Count of Participants; unit: Participants] — Patient institution data was pulled from INPC to database or supplied by caregivers who self-referred at events: Eskenazi, IU Health, or St. Vincent.
  Participants
    Eskenazi | 56 | 65 | 121
    IU Health | 42 | 37 | 79
    St. Vincent | 1 | 0 | 1
Functional Assessment Staging Tool for Dementia (FAST) [Number; unit: participants] — Caregivers responded "yes" or "no" to 12 questions regarding the functional ability of the person with dementia (PWD). Each question aligned with the stages in the FAST tool. Scoring calculated if PWD was stage 5 (moderate) through stages 6 (severe) and 7 (very severe).
  participants
    Moderate (FAST=5) | 4 | 4 | 8
    Severe (FAST=6-7) | 95 | 98 | 193
Patient Medical Conditions (Comorbidities) [Count of Participants; unit: Participants] — Caregivers responded "yes" or "no" if a doctor or another health care worker had diagnosed or treated the person with dementia (PWD) with the following medical problems in the past 3 years. Nine groups of medical issues were listed and a "yes" was counted if at least one item from a group was a "yes." Caregivers were instructed not to count the PWD Alzheimer's or dementia diagnosis as "another neurological condition" in the 6th item.
  Participants
    Asthma, emphysema, or chronic bronchitis: Yes | 18 | 11 | 29
    Asthma, emphysema, or chronic bronchitis: No | 81 | 91 | 172
    High blood pressure or hypertension: Yes | 71 | 73 | 144
    High blood pressure or hypertension: No | 28 | 29 | 57
    High blood sugar or diabetes: Yes | 25 | 29 | 54
    High blood sugar or diabetes: No | 74 | 73 | 147
    Arthritis or rheumatism (inflammation of the joints): Yes | 54 | 59 | 113
    Arthritis or rheumatism (inflammation of the joints): No | 45 | 43 | 88
    Angina, heart failure, or other types of heart disease: Yes | 33 | 36 | 69
    Angina, heart failure, or other types of heart disease: No | 66 | 66 | 132
    Stroke, seizures, Parkinson's disease, or another neurological condition: Yes | 25 | 37 | 62
    Stroke, seizures, Parkinson's disease, or another neurological condition: No | 74 | 65 | 139
    Liver disease: Yes | 2 | 2 | 4
    Liver disease: No | 97 | 100 | 197
    Kidney or renal disease: Yes | 16 | 18 | 34
    Kidney or renal disease: No | 83 | 84 | 167
    Cancer: Yes | 10 | 10 | 20
    Cancer: No | 89 | 92 | 181
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: score on a scale] — The MoCA was administered to support FAST stage screening results and caregiver self-report of the person with dementia's (PWD) cognitive decline. Scores for the MoCA range from 0-30 with 18-25 = mild cognitive impairment, 10-17= moderate cognitive impairment and less than 10= severe cognitive impairment. Population: The MoCA was administered with person with dementia (PWD) if caregiver gave permission. In some cases, the PWD was unable to take the test. When the IRB approved protocol amendment 12 to recruit fully remote and with verbal consent only, the MoCA was no longer administered during baseline.The total MoCAs administered for the study was 32.
  score on a scale
    number analyzed (Participants) | 16 | 16 | 32
    (all) | 10.5 (4.2) | 11.4 (4.5) | 10.9 (4.3)
Neuropsychiatric Inventory Questionnaire (NPI-Q: PWD) [Mean (Standard Deviation); unit: score on a scale] — The Neuropsychiatric Inventory Questionnaire measures the presence and severity of 12 neuropsychiatric symptoms in the person with dementia (PWD) in the past month per caregiver report. Each symptom reported as present is scored on a scale of 1-3 with higher scores indicating more severity of the symptom: mild, moderate, or severe. The NPI-Q Patient Symptom and Severity total score is constructed by summing the value of each presenting symptom's severity and ranges from 0-36 with higher scores indicating more severe patient neuropsychiatric symptoms.
  score on a scale | 9.9 (6.7) | 9.4 (6.4) | 9.7 (6.5)
Symptom Measures in End-of-Life Dementia (SM-EOLD) [Mean (Standard Deviation); unit: score on a scale] — The Symptom Measures in End-of-Life Dementia (SM-EOLD) measures the presence and frequency of 9 symptoms experienced by the person with dementia (PWD) in the previous 90 days per caregiver report: pain, shortness of breath, depression, fear, anxiety, agitation, calm, skin breakdown, and resistance to care. Each symptom is scored on a scale ranging from 0 to 5: never, once a month, 2 or 3 days a month, once a week, several days a week, daily. The SM-EOLD score is constructed by summing the value of each item, and ranges from 0-45 with higher scores indicating less symptom control (comfort).
  score on a scale | 29.8 (9) | 28.8 (8.8) | 29.3 (8.9)
Physical Self-Maintenance Scale/Activities of Daily Living (PSMS/ADLs) [Mean (Standard Deviation); unit: score on a scale] — The Physical Self-Maintenance Scale/Activities of Daily Living (PSMS/ADLs) measures the level of functioning of the person with dementia (PWD) in 6 basic and 7 instrumental ADLs in the previous 90 days per caregiver report. Only the 6 basic ADLs were included in analyses: toileting, bathing, dressing, grooming, physical ambulation, and feeding. Each ADL is scored as either 1 (independent in that activity) or 0 (needs assistance). The total score is constructed by summing the value of each of these 6 items and ranges from 0-6 with higher scores indicating less impairment and more independence.
  score on a scale | 1.1 (1.3) | 1.2 (1.5) | 1.1 (1.4)
Neuropsychiatric Inventory Questionnaire (NPI-Q: Caregiver Distress) [Mean (Standard Deviation); unit: score on a scale] — The Neuropsychiatric Inventory Questionnaire measures the presence and severity of 12 neuropsychiatric symptoms in the person with dementia (PWD) in the past month per caregiver report. If the symptom was reported as present, then the caregiver rated the level of distress they experienced related to the patient's symptom on a scale of 0-5 with higher scores indicating more distress. The NPI-Q Caregiver Distress total score is constructed by summing the value of each distress item and ranges from 0-60 with higher scores indicating more caregiver distress.
  score on a scale | 10.8 (9.2) | 10.4 (8.4) | 10.6 (8.8)
Patient Health Questionnaire (PHQ-8: Caregiver) [Mean (Standard Deviation); unit: score on a scale] — The Patient Health Questionnaire-8 item measures the frequency of depressive symptoms experienced by the caregiver in the last two weeks per caregiver report. Each symptom is scored on a scale of 0-3 (not at all, several days, more than half the days, nearly every day) with higher scores indicating more frequency of depressive symptoms. The PHQ-8 Caregiver total score is constructed by summing the value of each item and ranges from 0-24 with higher scores indicating more frequent depressive symptoms in the caregiver.
  score on a scale | 3.7 (4.2) | 4.1 (4) | 3.9 (4.1)
Caregiver Strain Index [Mean (Standard Deviation); unit: units on a scale] — The Caregiver Strain Index is a screening instrument which can be used to identify strain of carers, assess their ability to go on caring and to identify areas where support may be needed. Caregivers responded "yes" or "no" to 13 questions. The total score is determined by a count of the "Yes" answers. Scores may range from 0-13; a score of 7 or greater indicates a high level of stress.
  units on a scale | 6.6 (3.8) | 6.8 (3.5) | 6.7 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Neuropsychiatric Inventory Questionnaire (NPI-Q) for Patient Symptom and Severity
Description: The Neuropsychiatric Inventory Questionnaire measures the presence and severity of 12 neuropsychiatric symptoms in the person with dementia (PWD) in the past month per caregiver report. Each symptom reported as present is scored on a scale of 1-3 with higher scores indicating more severity of the symptom: mild, moderate, or severe. The NPI-Q Patient Symptom and Severity total score is constructed by summing the value of each presenting symptom's severity and ranges from 0-36 with higher scores indicating more severe patient neuropsychiatric symptoms.
Time Frame: 0-24 months
Population: This outcome measure was collected at baseline, 3, 6, 9 12, 15, 18, 21 and 24 months for each participant active on study at that time point and with a caregiver available to respond. The number entered represents the mean across all time points for both groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IN-PEACE Dementia Care Coordination | Usual Care
Number analyzed (Participants) | 99 | 102
score on a scale | 9.149 (0.747) | 9.39 (0.756)
Statistical Analysis 1: Comparison: IN-PEACE Dementia Care Coordination vs Usual Care; Test type: Superiority — Longitudinal measures of NPI-Q patient over 24 months were compared between the two groups using mixed effects model that included a group indicator variable, time since baseline, and an interaction between group and time as independent variables. Unstructured variance-covariance matrix was used to adjust for within-subject correlations over time. Predicted differences in mean scores between the two groups at each time point were estimated using the contrast procedures in the mixed model; p = 0.8719, Mixed Models Analysis

2. Secondary Outcome: Symptom Management - End of Life for Dementia (SM-EOLD)
Description: The Symptom Measures in End-of-Life Dementia (SM-EOLD) measures the presence and frequency of 9 symptoms experienced by the person with dementia (PWD) in the previous 90 days per caregiver report: pain, shortness of breath, depression, fear, anxiety, agitation, calm, skin breakdown, and resistance to care. Each symptom is scored on a scale ranging 0 - 5 (daily, several days a week, once a week, 2 or 3 days a month, once a month, never) with higher scores indicating better symptom control. The SM-EOLD total score is constructed by summing the value of each item, and ranges from 0-45 with higher scores indicating better symptom control (comfort).
Time Frame: 0-24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IN-PEACE Dementia Care Coordination | Usual Care
Number analyzed (Participants) | 99 | 102
score on a scale | 28.36 (0.972) | 26.133 (0.984)
Statistical Analysis 1: Comparison: IN-PEACE Dementia Care Coordination vs Usual Care; Test type: Superiority — Longitudinal measures of SM-EOLD over 24 months were compared between the two groups using mixed effects model that included a group indicator variable, time since baseline, and an interaction between group and time as independent variables. Unstructured variance-covariance matrix was used to adjust for within-subject correlations over time. Predicted differences in mean scores between the two groups at each time point were estimated using the contrast procedures in the mixed model; p = 0.8389, Mixed Models Analysis

3. Secondary Outcome: Patient Health Questionnaire (PHQ-8) Caregiver
Description: The Patient Health Questionnaire-8 item measures the frequency of depressive symptoms experienced by the caregiver in the last two weeks per caregiver report. Each symptom is scored on a scale of 0-3 (not at all, several days, more than half the days, nearly every day) with higher scores indicating more frequency of depressive symptoms. The PHQ-8 Caregiver total score is constructed by summing the value of each item and ranges from 0-24 with higher scores indicating more frequent depressive symptoms in the caregiver.
Time Frame: 0-24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IN-PEACE Dementia Care Coordination | Usual Care
Number analyzed (Participants) | 99 | 102
score on a scale | 4.472 (0.507) | 4.522 (0.511)
Statistical Analysis 1: Comparison: IN-PEACE Dementia Care Coordination vs Usual Care; Test type: Superiority — Longitudinal measures of PHQ-8 over 24 months were compared between the two groups using mixed effects model that included a group indicator variable, time since baseline, and an interaction between group and time as independent variables. Unstructured variance-covariance matrix was used to adjust for within-subject correlations over time. Predicted differences in mean scores between the two groups at each time point were estimated using the contrast procedures in the mixed model; p = 0.3431, Mixed Models Analysis

4. Secondary Outcome: Neuropsychiatric Inventory Questionnaire (NPI-Q) Caregiver Distress
Description: The Neuropsychiatric Inventory Questionnaire measures the presence and severity of 12 neuropsychiatric symptoms in the person with dementia (PWD) in the past month per caregiver report. If the symptom was reported as present, then the caregiver rated the level of distress they experienced related to the patient's symptom on a scale of 0-5 with higher scores indicating more distress. The NPI-Q Caregiver Distress total score is constructed by summing the value of each distress item and ranges from 0-60 with higher scores indicating more caregiver distress.
Time Frame: 0-24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IN-PEACE Dementia Care Coordination | Usual Care
Number analyzed (Participants) | 99 | 102
score on a scale | 9.282 (1.063) | 10.148 (1.073)
Statistical Analysis 1: Comparison: IN-PEACE Dementia Care Coordination vs Usual Care; Test type: Superiority — Longitudinal measures of NPI-Q caregiver distress over 24 months were compared between the two groups using mixed effects model including a group indicator variable, time since baseline, and an interaction between group and time as independent variables. Unstructured variance-covariance matrix was used to adjust for within-subject correlations over time. Predicted differences in mean scores between the two groups at each time point were estimated using the contrast procedures in the mixed model; p = 0.6612, Mixed Models Analysis

5. Secondary Outcome: Emergency Department Visits and Hospitalizations
Description: Combined measure of counts of emergency department (ED) visits and hospital admissions drawn from hospital reported data in the Indiana Network for Patient Care (INPC) database, managed by the Indiana Health Information Exchange (IHIE). As pre-specified, this data only includes the patient from each dyad and not the caregiver.
Time Frame: 0-24 months
Population: As pre-specified, this data only includes the patient from each dyad and not the caregiver.
Measure: Count of Participants; unit: Participants
Arm/Group | IN-PEACE Dementia Care Coordination | Usual Care
Number analyzed (Participants) | 99 | 102
Participants | 50 | 80
Statistical Analysis 1: Comparison: IN-PEACE Dementia Care Coordination vs Usual Care; Test type: Superiority — A zero-inflated Poisson (ZIP) model was used to compare the mean numbers of hospitalization/ED events between the two groups. The ZIP model consists of a combination of a standard Poisson distribution for count data and a binary logistic regression model to account for additional zero events exceeding what would be expected from an underlying Poisson distribution; p = 0.0007, Zero-Inflated Poisson Regression Model

ADVERSE EVENTS:
Time Frame: Through study completion, up to 24 months or the death of the patient
Description: Adverse events could be reported by caregivers during intervention visits and also were systematically collected for both arms every three months: death, emergency department visits, hospitalizations, falls, elopements, and other accidents. This data was collected only on the patients from each dyad as pre-specified; caregivers were not monitored nor assessed for mortality or adverse events. Death is an expected outcome for the patient population's condition under study.
Arm/Group | IN-PEACE Dementia Care Coordination | Usual Care
All-Cause Mortality (participants affected / at risk) | 40/99 | 43/102
Serious Adverse Events (participants affected / at risk) | 50/99 | 61/102
Other Adverse Events (participants affected / at risk) | 77/99 | 89/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IN-PEACE Dementia Care Coordination (N=99) | Usual Care (N=102)
Hospitalizations (General disorders) | 50 (82) | 61 (113)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IN-PEACE Dementia Care Coordination (N=99) | Usual Care (N=102)
Falls (Nervous system disorders) | 35 (70) | 42 (78)
Elopements (Nervous system disorders) | 26 (35) | 15 (19)
Other Accidents (General disorders) | 8 (12) | 7 (12)
ED Visits (General disorders) | 60 (125) | 81 (212)

LIMITATIONS AND CAVEATS:
Study subjects drawn primarily from two health systems in central Indiana and required to have an English-speaking caregiver. No technical difficulties; targeted enrollment completed on time and intervention and data collection very complete despite coronavirus disease 2019 (COVID-19) pandemic and move to fully remote operations. Low levels of symptoms in patients and caregivers in both arms may have limited ability to demonstrate impact of intervention on these measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT03773757/Prot_SAP_002.pdf
  • Informed Consent Form (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT03773757/ICF_000.pdf